CLINICAL TRIAL: NCT06968767
Title: Evaluation Of Preparation Time Of Bioflx Crowns Compared To Zirconia Crowns On Primary Molars
Brief Title: Preparation Time Of Bioflx Crowns Compared To Zirconia Crowns On Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Halah Mosaed Ali Alshaeri, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-BFC VS ZRC
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A performed bioflx crown (Experimental): (Nu smile, united state) introduced Biofix Crowns and claimed as the first flexible, durable, and esthetic preformed crown for primary molars. Biofix Crowns are monochromatic, metal-free, tooth-colored crowns made up of high-strength resin polymer used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are like SSC in tooth preparation as claimed by the manufacturer. Their flexibility and snap-fit technology aim to improve retention while minimizing trauma during placement.
  Interventions: Other: bioflx crown
- group B performed zirconia crown (Experimental): NuSmile Zirconia Crowns are prefabricated, esthetic full-coverage restorations designed for primary teeth. Known for their superior strength, durability, and natural tooth-like appearance, these crowns provide an excellent alternative to traditional stainless steel crowns. Made from high-quality medical-grade zirconia, they are biocompatible, resistant to chipping, and highly polished to minimize plaque accumulation and gingival irritation.
  NuSmile Zirconia Crowns require significant tooth preparation for proper fit and retention. They are available in various sizes to accommodate different primary molars and anterior teeth. Their lifelike translucency and color-matching capabilities make them a preferred choice for parents and clinicians.
  Interventions: Other: zirconia crown

INTERVENTIONS:
Other: bioflx crown — (Group A: Preformed Biofix Crown - Assigned Intervention)
  Crown Selection & Tooth Preparation:
  Measure the mesiodistal width using calipers to select an appropriately sized crown. If a mesial or distal wall is missing, use the contralateral tooth for size selection. Choose the crown that closely matches the measured mesiodistal width. Select the smallest crown that preserves proximal contacts using a trial-and-error approach. If crimping is necessary, use Howe's pliers.
  Perform 1-1.5 mm occlusal reduction using a tapered diamond bur.
  Reduce proximal areas by approximately 0.5 mm to clear the contact area.
  Crown Placement & Cementation:
  Ensure a snug fit of the selected crown. Apply a thin layer of glass ionomer cement inside the crown. Seat the crown firmly using finger pressure. Have the child bite down gently to ensure proper seating.
  Final Adjustments & Cleanup:
  Remove excess cement with floss or an explorer. Verify the crown's fit, occlusion, and stability.
  Arms: group A performed bioflx crown
Other: zirconia crown — Group B: Preformed Zirconia Crown - Assigned Intervention)
  Crown Selection:
  Measure the mesiodistal width using calipers to select the appropriate crown. If a mesial or distal wall is missing, use the contralateral tooth for size selection. Choose the one that closely matches the mesiodistal width. Select the smallest crown that preserves proximal contacts.
  Tooth Preparation:
  Reduce the occlusal surface by 1.5-2 mm using a tapered diamond bur.
  Reduce interproximal areas by 1-1.5 mm, ensuring a feather-edge finish.
  Perform a 1-2 mm subgingival preparation in passively placed fissure bur.
  Crown Placement & Passive Fit Check:
  Place the selected crown on the prepared tooth.
  Cementation of the Crown:
  Apply a thin layer of glass ionomer cement inside the crown. Seat the crown with passive finger pressure. Have the child bite down gently to ensure seating.
  Arms: group B performed zirconia crown

SUMMARY:
This study aims to evaluate and compare the preparation time required for Bioflx crowns versus zirconia crowns on primary molars through a randomized clinical trial.

• Primary Objective: To compare the preparation time required for Bioflex crowns and zirconia crowns on primary molars in pediatric patients.

• Secondary Objectives:

To evaluate the clinical performance of Bioflex crowns compared to zirconia crowns, including:

Retention, Patient Satisfaction, Parental Satisfaction, Occlusal Wear and Gingival Health.

the main question it aim to answer: Is there a significant difference in the preparation time required for Bioflx crowns compared to zirconia crowns in the primary molars of pediatric patients?

DETAILED DESCRIPTION:
In pediatric dentistry, achieving efficient and aesthetic restoration of primary molars remains a significant challenge, particularly when treating young or anxious patients who may struggle with long or complex procedures. Zirconia crowns are widely used due to their durability, excellent biocompatibility, and natural tooth-like appearance, making them the gold standard for full-coverage aesthetic restorations in children. However, their placement involves extensive tooth preparation, which results in longer chair time and an increased risk of pulp exposure. These factors can negatively impact both treatment outcomes and patient behavior management.

Bioflex crowns have emerged as a potential alternative, offering a more flexible and user-friendly design that simplifies placement and reduces the amount of tooth preparation required. This may result in shorter procedure times and improved patient comfort. Despite these potential benefits, there is currently limited clinical evidence comparing the preparation time and efficiency of Bioflex crowns versus zirconia crowns for restoring primary molars.

This gap in knowledge makes it difficult for clinicians to make fully informed decisions about which crown system offers the best balance of procedural efficiency, aesthetics, and patient cooperation. By directly comparing Bioflex and zirconia crowns in terms of tooth preparation time and overall clinical practicality, the proposed study aims to determine whether Bioflex crowns provide a significant advantage in pediatric settings. The results could help identify the most time-efficient and effective restorative option for primary molars, ultimately improving care outcomes for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 8 years with a primary molar that needs to be covered by a crown.

Medically healthy children (ASA I or II according to the American Society of Anesthesiologists classification).

Children whose parent or guardian is willing to sign an informed consent.

Children whose parent or guardian are willing to comply with follow-up visits.

Frankl's positive and definitely positive patient.

Exclusion Criteria:

* Molars with severe structural loss that may compromise crown retention.

Children with poor oral hygiene that may contribute to higher plaque levels and affect the clinical outcomes of the crown restorations.

Children with a history of allergies; known allergies to dental local anesthesia or to the materials used in Biofix crowns.

Children with any systemic conditions or disabilities that may affect their ability to participate in the study.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
prepration time | time frame: T0: 0 basline, follow up 12 month
  measured by stop watch per minutes

SECONDARY OUTCOMES:
Occlusal wear of crown | T (Time): 12 months Intervals: T0: 0, T1: 3 months, T2: 6 months, T3: 12 months
  Measure: By Modified United States Public Health System criteria
  Criteria:
  Alpha: Occlusal surface intact
  Bravo: Wear of occlusal surface without tooth surface exposure
  Charlie: Wear of occlusal surface with exposure
  Measure: By Modified United States Public Health System criteria
  Criteria:
  Alpha: Occlusal surface intact
  Bravo: Wear of occlusal surface without tooth surface exposure
  Charlie: Wear of occlusal surface with exposure
  Measure: By Modified United States Public Health System criteria
  Criteria:
  Alpha: Occlusal surface intact
  Bravo: Wear of occlusal surface without tooth surface exposure
  Charlie: Wear of occlusal surface with exposure
retention | Follow-up: 12 months Intervals: T0: 0, T1: 3 months, T2: 6 months, T3: 12 months
  Measure: By Modified United States Public Health System criteria
  Criteria:
  Alpha: Intact
  Bravo: Chipped/loss of material
  Charlie: Complete loss of crown
Gingival Health | 12 months Intervals: T0: 0, T1: 3 months, T2: 6 months, T3: 12 months
  Measure: By Gingival Index
  Scores:
  0: Healthy gum
  1. Mild inflammation and edematous gingiva, no bleeding on probing
  2. Red edematous and shiny gingiva, bleeding on probing
  3. Red edematous and ulcerated gingiva, spontaneous bleeding
Child and parental satisfaction | T (Time): 12 months Intervals: T0: 0, T1: 3 months, T2: 6 months, T3: 12 months
  Measure: By 5-point Likert scale (Units of measurement)
  1. Very happy
  2. Happy
  3. Neither
  4. Unhappy
  5. Very unhappy Questionnaire Type: Ordinary or N/A (Existing validated tool)

CONTACTS AND LOCATIONS:
Overall Officials: Hala m Alshaeri, Bachelor of Dental surgery, Principal Investigator — Cairo university faculty of dentistry
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38911945/